CLINICAL TRIAL: NCT03740607
Title: Virtual Reality for Alleviation of Peripheral IV Placement-Associated Discomfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Annie Chow, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: c.2017.114d
Record Dates: First submitted 2018-11-10; First posted 2018-11-14 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Procedural Anxiety; Procedural Pain; Perioperative Care
Keywords: Adult; Peripheral IV; procedural pain; procedural anxiety; virtual reality; peripheral intravenous catheter
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: randomized prospective cohort
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Virtual reality during PIV placement (Experimental): Randomized consented adult subjects will participate in a six-minute healthcare virtual reality software program via Samsung Gear virtual reality headsets while receiving 18 or 20-gauge peripheral intravenous catheter placement in peri-operative suite in preparation for surgery. They will be asked to rate their pain and discomfort afterwards using a graphic rating scale. They will be asked several questions about satisfaction, in order to elicit clinical significance of this intervention. Demographic information will be collected, and baseline vital signs upon arrival to OR will be abstracted retrospectively.
  Interventions: Device: Virtual reality; Procedure: Peripheral intravenous catheter placement
- Standard PIV placement (Placebo Comparator): Adult control arm subjects will receive 18 or 20-gauge peripheral intravenous catheter placement according to current standard protocol, without virtual reality distraction .They will be asked to rate pain and discomfort afterwards using a graphic rating scale. Demographic information will be collected, and baseline vital signs upon arrival to OR will be abstracted retrospectively.
  Interventions: Procedure: Peripheral intravenous catheter placement

INTERVENTIONS:
Device: Virtual reality — Healthcare virtual reality software implemented during peripheral intravenous catheter placement
  Other Names: Samsung Gear Headset, AppliedVR software
  Arms: Virtual reality during PIV placement
Procedure: Peripheral intravenous catheter placement — Peripheral intravenous catheters are placed in the peri-operative suites in preparation for anesthesia during surgery.
  Other Names: IV; PIV

SUMMARY:
Immersive virtual reality (iVR) has been used successfully to manage pain with distraction. It is a non-invasive treatment modality unassociated with worrisome well-known side effects typically seen when opioids and NSAIDS are used, and has previously been used safely in place of analgesia during dressing changes and burn care. This study investigates whether iVR can be useful as a stand-alone option to manage the pain associated with placement of peripheral intravenous (PIV) catheters in adults.

DETAILED DESCRIPTION:
This is a prospective study of the effect of immersive virtual reality on the perception of pain during peripheral IV (PIV) placement. Adult patients who require PIV placement for elective surgery will be consented for intervention while in the peri-operative suites (PS). The VR intervention will consist of a headset and immersive VR software that allows the patient to engage in a virtual world during PIV placement. Subjects will be queried immediately after PIV placement using the validated graphic rating scale regarding the sensory, cognitive, and affective aspects of discomfort they experienced with PIV placement (Appendix A). They will also be asked two validated questions concerning patient satisfaction (Dexter et al 1997). A control group of patients will undergo a similar assessment with slightly different wording after receiving PIV placement without iVR.

ELIGIBILITY:
Inclusion Criteria:

Brooke Army Medical Center patients age 19-89 undergoing peripheral intravenous catheter placement in preparation for elective surgery will be eligible for participation.

Exclusion Criteria:

Patients will be excluded with head wounds/head bandages preventing the use of a headset, active nausea/vomiting, history of seizure, dementia, psychosis, mania, vertigo, or motion sickness, if the patient is pregnant or incarcerated on the day of surgery, and if the patient is unable to consent self.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Discomfort associated with peripheral IV placement | This outcome will be measured immediately after peripheral IV placement
  Subject experiences will be measured using a validated graphic rating scale (GRS) which enquires about the extent to which the experience was unpleasant.

SECONDARY OUTCOMES:
Magnitude of pain severity | This outcome will be measured immediately after peripheral IV placement
  Subjects will rate their worst pain during the IV placement on a scale of 1-10 out of 10 possible points
Time spent thinking about pain | This outcome will be measured immediately after peripheral IV placement
  Subject will describe the amount of time spent thinking about pain during IV placement, as a proportion.
Degree to which subject felt immersed in virtual reality | This outcome will be measured immediately after peripheral IV placement
  The subject will answer a question regarding the extent to which they felt they went "inside" the computer-generated world
Nausea | This outcome will be measured immediately after peripheral IV placement
  Subject will answer a question regarding extent to which nausea was experienced during IV placement
Claustrophobia | This outcome will be measured immediately after peripheral IV placement
  The subject will be asked to answer a question about the extent to which they felt claustrophobic for any reason during IV placement
Clinical significance | This outcome will be measured immediately after peripheral IV placement
  the subject will be asked if they would want to have their IV placed this way again
Satisfaction score | This outcome will be measured immediately after peripheral IV placement
  The subject will be asked if they were satisfied with IV placement
Physiological parameters | Initial vital signs at start of anesthesia care will be abstracted retrospectively. This reading will likely occur within an hour of the initial intervention, as start times for anesthesia cases are within an hour of initiation of peri-operative care
  Baseline vital signs- continuous variables
Fun factor | This outcome will be measured immediately after peripheral IV placement
  Subject will describe the extent to which they found the experience to be fun, on a scale of 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Maani, MD, Study Director — BAMC Faculty
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maani CV, Hoffman HG, Fowler M, Maiers AJ, Gaylord KM, Desocio PA. Combining ketamine and virtual reality pain control during severe burn wound care: one military and one civilian patient. Pain Med. 2011 Apr;12(4):673-8. doi: 10.1111/j.1526-4637.2011.01091.x. Epub 2011 Apr 11. PMID 21481162
- [Background] Maani CV, Hoffman HG, Morrow M, Maiers A, Gaylord K, McGhee LL, DeSocio PA. Virtual reality pain control during burn wound debridement of combat-related burn injuries using robot-like arm mounted VR goggles. J Trauma. 2011 Jul;71(1 Suppl):S125-30. doi: 10.1097/TA.0b013e31822192e2. PMID 21795888
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Background] Rosen LD, Whaling K, Carrier LM, Cheever NA, Rokkum J. The Media and Technology Usage and Attitudes Scale: An empirical investigation. Comput Human Behav. 2013 Nov 1;29(6):2501-2511. doi: 10.1016/j.chb.2013.06.006. PMID 25722534
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Hoffman HG, Richards TL, Van Oostrom T, Coda BA, Jensen MP, Blough DK, Sharar SR. The analgesic effects of opioids and immersive virtual reality distraction: evidence from subjective and functional brain imaging assessments. Anesth Analg. 2007 Dec;105(6):1776-83, table of contents. doi: 10.1213/01.ane.0000270205.45146.db. PMID 18042882
- [Background] Hoffman HG, Patterson DR, Seibel E, Soltani M, Jewett-Leahy L, Sharar SR. Virtual reality pain control during burn wound debridement in the hydrotank. Clin J Pain. 2008 May;24(4):299-304. doi: 10.1097/AJP.0b013e318164d2cc. PMID 18427228
- [Background] Dexter F, Aker J, Wright WA. Development of a measure of patient satisfaction with monitored anesthesia care: the Iowa Satisfaction with Anesthesia Scale. Anesthesiology. 1997 Oct;87(4):865-73. doi: 10.1097/00000542-199710000-00021. PMID 9357889
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523
- [Background] Kenney MP, Milling LS. The effectiveness of virtual reality distraction for reducing pain: a meta-analysis. Psychology of Consciousness: Theory, Research, and Practice 3(3): 199-210, 2016.